CLINICAL TRIAL: NCT02180282
Title: Impact of the M22-IPL Acne Filter on Acne Vulgaris
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruiting rate
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-M22-IPL-14-01
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Acne
Keywords: Acne Treatment
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acne Treatment (Experimental): Acne treatment using the M22-IPL acne filter
  Interventions: Device: M22-IPL

INTERVENTIONS:
Device: M22-IPL — The M22 is an advanced computer-controlled light emission system that incorporates several different light modules.
  The IPL hand piece operates at a spectrum of 400-1200nm with 7 different filters that can be easily inserted to the hand piece to treat different conditions. The IPL hand piece also includes 2 different sapphire cooled light guides of 8x15mm and 15x35mm. The cut-off filter that will be used for this evaluation is the Acne Filter that cuts off all light with the wavelength of 400-600 and 800-1200nm.

SUMMARY:
Up to 20 healthy subjects age 15-45 years old ,Skin Phototype I-V,Study will be conducted in 1 site.

Primary objectives is to evaluate the efficacy of IPL acne filter treatment for improvement of acne vulgaris as assessed by lesion count.

.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and provide written Informed Consent;
2. Healthy male or female, 15-45 years of age;
3. Fitzpatrick skin type I-V;
4. Have at least 15 inflammatory lesions (papules and pustules) in the face.
5. Having clinical diagnosis of mild to moderate inflammatory acne on face with Investigator Global Acne scale = 2 and 3;
6. Able and willing to comply with the treatment/follow-up schedule and requirements;
7. Women of child-bearing age are required to be using a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, Nova ring, and partner with vasectomy or abstinence) at least 3 months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

1. Skin type VI;
2. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding;
3. Heavy smoker (>1 pack of cigarettes a day);
4. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study;
5. Photosensitivity or any sensitivity to the sun that causes a rash or allergic reaction;
6. Use of photosensitive medication for which light exposure is contraindicated;
7. Treatment with topical retinoid therapy or antibiotics for the treatment of acne within 2 weeks of study enrollment or during the study.
8. Treatment with oral retinoid medications (Accutane® or Soriatane®) within 6 months of the study enrollment or during the study.
9. Treatment with any topical or systemic anti acne therapy for at least 2 weeks prior to starting the study treatment or during the study.
10. Any history of gold therapy;
11. Prior use of collagen, fat injections or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 12 months of initial treatment or during the course of the study. Treatment may not be performed at all over permanent dermal implants;
12. Prior ablative resurfacing procedure or face lift in treated area with laser or other devices within 12 months of initial treatment or during the course of the study;
13. Any other surgery in treated area within 9 months of initial treatment or during the course of the study;
14. Participation in a study of another investigational device or drug involving the same anatomical site within 3 month prior to enrollment or during this evaluation, or if not involving the same anatomical site, as per the Investigator's discretion;
15. History of keloid or any other type of hypertrophic scar formation or poor wound healing in a previously injured skin area;
16. Showing symptoms of hormonal disorders, as per the Investigator's discretion (such as Melasma, Chloasma);
17. Concurrent inflammatory skin conditions, Open laceration or abrasion of any sort on area to be treated during the course of treatment;
18. Active Herpes Simplex at the time of treatment or having experienced more than three episodes of Herpes Simplex eruption within a year of study enrollment;
19. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to each treatment (as per the patient's physician discretion);
20. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications;
21. Having any form of active cancer at the time of enrollment and during the course of the study or history of skin cancer on the face;
22. Mentally incompetent or evidence of active substance or alcohol abuse;
23. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study;
24. For subjects undergoing test spots: considerable undesired response consisting of skin hypopigmentation (long term whitening), a scar or pre scar formation or any response deemed by the Investigator as grounds for exclusion.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
lesion count of acne vulgaris will be reduced by at least 50% for >75% of the study population. | week 6 (week 1 after the last treatment)
  The numbers of lesions are counted on each side of the face according to lesion type

SECONDARY OUTCOMES:
Investigator Global Assessment (IGA) Scale for Acne Vulgaris | following the treatments: at Baseline ,5 weeks and at follow up 6 and 10 weeks.
  The investigator will be required to grade the acne severity using the IGA scale
Subject Discomfort Evaluation | Following the treatments: Baseline,2,3,4,5 weeks
  Subject assessment of pain and discomfort associated with treatments using a Pain Visual Analogue Scale (VAS), were 0 is "no pain" and 100 is "intolerable pain.
Long term side effect and adverse events | throughout the duration of the study (Baseline,2,3,4,5 weeks)
  Any adverse events associated with various setting used during the treatment and follow-up period
Subject Downtime Evaluation | Following treatments baseline,2,3,4,5 weeks
  The downtime will be defined as the period of time following the procedure during which the subject had edema and erythema and felt unable/unwilling to go out in public
Subject Satisfaction | week 4 ,6 ,10
  The assessment will be based on a 5-point Likert scale detailed in Table 5 where 0 represents dissatisfied and 4 represents very satisfied.
The Cardiff Acne Disability Index | Baseline ,4,6,10 weeks
  The Cardiff Acne Disability Index is a short 5 item questionnaire derived from the longer Acne Disability Index
Subject personal experience | week 10
  Subject's likelihood of recommending the treatment or seeking additional treatments recorded in a questionnaire using a six point scale: 1=Extremely Unlikely; 2=Very Unlikely; 3=Somewhat Unlikely; 4=Somewhat likely; 5=Very likely; 6=Extremely likely

CONTACTS AND LOCATIONS:
Overall Officials: Dr. J. Matthew Knight, MD, FAAD, Principal Investigator — Knight Dermatology Institute
Locations (1):
- Knight Dermatology Institute, Orlando, Florida, United States